CLINICAL TRIAL: NCT06909916
Title: Assessment of Bone Displacement Under Loading Following Distal Femur Periprosthetic Fracture Repair With Weight-Bearing CT and Conventional CT
Brief Title: Weight-Bearing CT and Conventional Periprosthetic Distal Knee Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14154
Record Dates: First submitted 2024-08-06; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-08

CONDITIONS: Periprosthetic Fracture Around Prosthetic Joint Implant

STUDY DESIGN:
Intervention Model Description: One single visit: 1 loaded and 2 unloaded scans with weight-bearing CT. One loaded and 2 unloaded scans with conventional CT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Periprosthetic Fracture Knee Repaired (Experimental): The one and only group will be participants that have undergone revision surgery for at least 1> year prior for their periprosthetic distal knee fracture.
  Interventions: Other: Periprosthetic Fracture Knee Repaired CT Scans

INTERVENTIONS:
Other: Periprosthetic Fracture Knee Repaired CT Scans — The investigators will be assessing the use of weight-bearing CT and conventional CT, specifically its imaging, with RSA-like software, for analyzing fracture healing for a periprosthetic distal knee fracture.

SUMMARY:
Total knee arthroplasty (TKA) is a surgical procedure commonly conducted for patients with end-stage knee osteoarthritis, often leading to improved pain relief and function. However, for patients that have suffered an associated periprosthetic fracture, a broken bone that occurs around the implant of a TKA, they may receive sub-optical care due to a lack of a trustworthy assessments for component fixation and fracture healing in the literature. The prevalence of TKA surgeries is increasing annually and is projected to rise further due to an ageing population and obesity issue. By extension to this primary surgery, more Canadians will require an invasive revision surgery that risks patient morbidity and mortality. Thus, it is imperative to set a standard for fixation and bone healing assessments to lessen revision burdens and improve patient outcomes. CT imaging can effectively visualize areas of incomplete bone ingrowth that may be hidden from overlapping anatomy on plain radiographs, which remains the go-to imaging modality for orthopaedic surgeons to assess periprosthetic fracture healing. The purpose of this prospective cross-sectional study is to examine the efficacy of weight-bearing CT as a diagnostic tool for 20 participants who experienced a distal femur periprosthetic fracture and underwent revision surgery using a fracture fixation plate and screws. Participants will be scanned under loaded and unloaded conditions. Radiographic outcomes will be evaluated, including bone segment displacement and its relation to participants' reports of pain.

DETAILED DESCRIPTION:
Total knee arthroplasty is the most cost-effective and successful treatment for knee joints with end-stage osteoarthritis, with more than 58,000 TKA surgeries in Canada in 2021-2022.1 The prevalence of TKA surgeries is increasing per year and is projected to rise due to an ageing population and obesity problems.1 In addition to the primary surgery, more than 4,000 Canadians require revision TKA surgery per year; the TKA revision burden is estimated to reach $13 billion by 2030 as a consequence of a substantial increase of 149% in primary surgeries by 2030 in the United States.1-3 Revision surgery is more invasive than primary surgery and poses the risk of increasing patient mortality rates, especially for older adults.3 Thus, it is imperative for surgeons to make an appropriate radiographic diagnosis of implant fixation and/or fracture healing, but many cases remain challenging to diagnose.4

In the orthopaedic literature, there is no consensus on a reliable definition criterion for long-bone non-unions, making the standardization of diagnoses difficult; the lack of a trustworthy assessment for component fixation and fracture healing can lead to patients receiving sub-optimal care.5 This can also limit the collection of evidence supporting the use of specific implant components, surgical techniques, and post-operative activity guidelines. Moreover, comparing healing results of different clinical studies for long-bone non-unions can become problematic due to different criteria being used.5 Radiographic features associated with loosening such as radiolucencies are often only appreciable for the cement-bone interface, rather than the cement-implant interface which is the most common site of failure causing loosening.4 Failure to properly diagnose fracture non-union leaves patients in pain with substantial morbidity, while unnecessary surgery risks significant complication. Given the increasing rates of TKA and associated predictions of increasing revision burden,6 along with ongoing debates over the superiority of certain implants or surgical techniques, there is an unmet need for better fixation and bone healing assessment.

Historically, radiostereometric analysis (RSA) has been the gold standard for measuring implant fixation.7 However, it remains a niche tool limited to clinical research because of its requirement for implanted marker beads and specialized equipment being accessible for a handful of labs in North America.7-8 Recently, multiple groups have developed approaches to perform RSA-like measurements using clinical CT scans for shoulder, hip, and knee replacements.9 The accuracy and precision of the "CT-RSA" methods are on par with conventional RSA and acceptable for clinical studies.10-15 It is predicted that there will be a greater uptake of CT-RSA than conventional RSA, but the technology is still in its infancy.9 The application of CT-RSA will undoubtedly be more inclusive as examinations can now be performed on patients who did not have marker beads implanted at the time of their original surgery, and CAD models of implants are not needed.16

Using a weight-bearing CT scanner is the most similar implementation of CT-RSA to conventional RSA, as exams can be acquired in unloaded and loaded positions. However, the availability of weight- bearing CT will always be lesser than conventional clinical CT scanners, even as more and more high volume orthopaedic centres are acquiring weight-bearing CT scanners. While some groups have implemented specialized loading devices to perform such scans with conventional CT,17 a more generalizable approach of simple internal-external leg rotations held in place with tape would ultimately offer the greatest potential uptake across centres.

The results of this proposed study will demonstrate the ability to precisely measure displacements between bone segments under loading following periprosthetic fracture repair with weight-bearing CT and conventional CT scanners. These will be the first-ever measurements of distal femur periprosthetic fracture healing with weight-bearing CT-RSA. Demonstration of this will enable us to pursue future studies that are prospective in nature and may evaluate topics such as time to weight-bearing activities, different types of surgical reconstructions, and relationship between healing and bone quality/bone health. Other centres with access to weight-bearing CT will also benefit from this work. Consideration for the ability to perform similar measurements with conventional CT in place of weight-bearing CT will improve the generalizability of this approach and support it as a clinical diagnostic tool. For example, surgeons may better understand bone fragment motion over time and recommend appropriate postoperative activities for patients' weight-bearing tolerance. Therefore, the proposed study design will evaluate the ability to perform inducible displacement measurements following the surgical repair of distal femur periprosthetic fractures using both weight-bearing CT and conventional CT.

ELIGIBILITY:
Inclusion Criteria:

* Underwent revision surgery for repair of a distal femur fracture surrounding a primary TKA femoral component using a fracture fixation plate >1 year
* Age 50-90 years
* Body mass index up to 40kg/m2
* Able to provide informed consent
* Able and willing to do study assessments and follow instructions

Exclusion Criteria:

* Does not understand English
* Undergone revision surgery for any other indication
* Received Intramedullary nail or distal femur replacement
* Cannot independently stand on one leg in the weight-bearing CT during the inducible displacement exam

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Maximum Total Point Motion of Fracture Segments from Conventional CT scans | 1 visit is only required for which the outcome measure will then be assessed. Through study completion, approximately of 1 year.
  Weight-Bearing CT scans of participants will be analyzed for any potential movement between the fracture segments from the identified fracture lines. This will be reported as the maximum total point motion, which refers to the largest observed movement of a point along the fracture line from its initial position.
Maximum Total Point Motion of Fracture Segments from Conventional CT scans | 1 visit is only required for which the outcome measure will then be assessed. Through study completion, approximately of 1 year.
  Conventional CT scans of participants will be analyzed for any potential movement between the fracture segments from the identified fracture lines. This will be reported as the maximum total point motion, which refers to the largest observed movement of a point along the fracture line from its initial position.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) Questionnaire | 1 visit is only required for which the outcome measure will then be assessed. Through study completion, approximately of 1 year.
  This Pain and function questionnaire will be used to assess the pain and ability-to-function of the knee of the participant. This is a participant-reported outcome and it will be compared to the weight-bearing and conventional CT scans.
The Knee Society Score (KSS) Questionnaire | 1 visit is only required for which the outcome measure will then be assessed. Through study completion, approximately of 1 year.
  Knee function and patient outcome questionnaire that will be used to assess the pain and functionality of the knee of the participant. This is a participant-reported outcome and ut will be compared to the weight-bearing and conventional CT scans.
UCLA Activity Score Guideline Questionnaire | 1 visit is only required for which the outcome measure will then be assessed. Through study completion, approximately of 1 year.
  A questionnaire assessing physical activity level from 1 (low) to 10 (high) in patients. It will be used to assess the functionality of the knee of the participant. This is a participant-reported outcome and it will be compared to the weight-bearing and conventional CT scans.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Teeter, PhD, Study Director — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; Brent Lanting, MD, Principal Investigator — Lawson Health Sciences Centre; Lyndsay Somerville, PhD, Study Chair — London Health Sciences Centre; Patrick J Mixa, MD, Study Chair — Western University; James Howard, MD, Study Chair — London Health Sciences Centre
Locations (1):
- University Hospital - London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steele JR, Ryan SP, Jiranek WA, Wellman SS, Bolognesi MP, Seyler TM. Cost of Aseptic Revision Total Knee Arthroplasty at a Tertiary Medical Center. J Arthroplasty. 2021 May;36(5):1729-1733. doi: 10.1016/j.arth.2020.11.028. Epub 2020 Dec 17. PMID 33390337
- [Background] Sinclair ST, Orr MN, Rothfusz CA, Klika AK, McLaughlin JP, Piuzzi NS. Understanding the 30-day mortality burden after revision total knee arthroplasty. Arthroplast Today. 2021 Oct 4;11:205-211. doi: 10.1016/j.artd.2021.08.019. eCollection 2021 Oct. PMID 34660865
- [Background] Crellin CT, Pennings JS, Engstrom SM, Shinar AA, Polkowski GG, Martin JR. Aseptic tibial loosening: Radiographic identification remains a diagnostic dilemma. Journal of Orthopaedic Reports. 2023;2(4):100194. doi:10.1016/j.jorep.2023.100194
- [Background] Wittauer M, Burch MA, McNally M, Vandendriessche T, Clauss M, Della Rocca GJ, Giannoudis PV, Metsemakers WJ, Morgenstern M. Definition of long-bone nonunion: A scoping review of prospective clinical trials to evaluate current practice. Injury. 2021 Nov;52(11):3200-3205. doi: 10.1016/j.injury.2021.09.008. Epub 2021 Sep 10. PMID 34531088
- [Background] Klug A, Gramlich Y, Rudert M, Drees P, Hoffmann R, Weissenberger M, Kutzner KP. The projected volume of primary and revision total knee arthroplasty will place an immense burden on future health care systems over the next 30 years. Knee Surg Sports Traumatol Arthrosc. 2021 Oct;29(10):3287-3298. doi: 10.1007/s00167-020-06154-7. Epub 2020 Jul 15. PMID 32671435
- [Background] Aspinall GA, Dunbar MJ. Assessing clinical results and outcome measures. Surgical Treatment of Hip Arhtritis. 2009;30-36. Doi:10.1016/B978-1-4160-5898-4.00004-5
- [Background] Valstar ER, Gill R, Ryd L, Flivik G, Borlin N, Karrholm J. Guidelines for standardization of radiostereometry (RSA) of implants. Acta Orthop. 2005 Aug;76(4):563-72. doi: 10.1080/17453670510041574. PMID 16195075
- [Background] Rohrl SM. "Great balls on fire:" known algorithm with a new instrument? Acta Orthop. 2020 Dec;91(6):621-623. doi: 10.1080/17453674.2020.1840029. Epub 2020 Nov 4. No abstract available. PMID 33143497
- [Background] Angelomenos V, Mohaddes M, Itayem R, Shareghi B. Precision of low-dose CT-based micromotion analysis technique for the assessment of early acetabular cup migration compared with gold standard RSA: a prospective study of 30 patients up to 1 year. Acta Orthop. 2022 Apr 22;93:459-465. doi: 10.2340/17453674.2022.2528. PMID 35478261
- [Background] Broden C, Sandberg O, Olivecrona H, Emery R, Skoldenberg O. Precision of CT-based micromotion analysis is comparable to radiostereometry for early migration measurements in cemented acetabular cups. Acta Orthop. 2021 Aug;92(4):419-423. doi: 10.1080/17453674.2021.1906082. Epub 2021 Apr 6. PMID 33821746
- [Background] Stigbrand H, Brown K, Olivecrona H, Ullmark G. Implant migration and bone mineral density measured simultaneously by low-dose CT scans: a 2-year study on 17 acetabular revisions with impaction bone grafting. Acta Orthop. 2020 Oct;91(5):571-575. doi: 10.1080/17453674.2020.1769295. Epub 2020 May 26. PMID 32452289
- [Background] Eriksson T, Maguire GQ Jr, Noz ME, Zeleznik MP, Olivecrona H, Shalabi A, Hanni M. Are low-dose CT scans a satisfactory substitute for stereoradiographs for migration studies? A preclinical test of low-dose CT scanning protocols and their application in a pilot patient. Acta Radiol. 2019 Dec;60(12):1643-1652. doi: 10.1177/0284185119844166. Epub 2019 May 1. No abstract available. PMID 31042065
- [Background] Sandberg OH, Karrholm J, Olivecrona H, Rohrl SM, Skoldenberg OG, Broden C. Computed tomography-based radiostereometric analysis in orthopedic research: practical guidelines. Acta Orthop. 2023 Jul 20;94:373-378. doi: 10.2340/17453674.2023.15337. PMID 37493579
- [Background] Kievit AJ, Buijs GS, Dobbe JGG, Ter Wee A, Kerkhoffs GMMJ, Streekstra GJ, Schafroth MU, Blankevoort L. Promising results of an non-invasive measurement of knee implant loosening using a loading device, CT-scans and 3D image analysis. Clin Biomech (Bristol). 2023 Apr;104:105930. doi: 10.1016/j.clinbiomech.2023.105930. Epub 2023 Mar 3. PMID 36906985
- See also: Canadian Joint Replacement Registry — https://www.cihi.ca/sites/default/files/document/hip-knee-replacements-in-canada-cjrr-annual-report-2021-2022-en.pdf